CLINICAL TRIAL: NCT03577600
Title: Study in Children With Brain Tumors in Terminal Stages Using Advanced Functional Magnetic Resonance Imaging in a Compassionate Palliative Care Setting, With Quantum Magnetic Resonance Therapy (QMRT).
Brief Title: Compassionate Treatment in Children With Brain Tumors With the Cytotron®
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: suspended due to administrative problems
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Eduardo Javier Barragán Pérez, Chief of Neurology Department, Hospital Infantil de Mexico Federico Gomez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIM 2018-007
Record Dates: First submitted 2018-06-12; First posted 2018-07-05 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Pediatric Brain Tumor
Keywords: Recurrent Ependymoma; Brainstem Gliomas; Rotational Field Quantum Magnetic Resonance (RFQMR); Cytotron®; High Grade Gliomas; Quantum Magnetic Resonance Therapy (QMRT); Brain Tumor Recurrence
MeSH Terms: conditions — Ependymoma

STUDY DESIGN:
Intervention Model Description: A case-study study. The controls will be historical and 2 controls will be taken that will be matched to the age range (preschool, school age, early adolescent, late adolescent), type of tumor and location (infra or supratentorial). This study is expected to last for approximately 12 months, comprised of 4-8 weeks of enrollment period, 28 days of treatment and 6 months of follow up. The enrollment will be completed prior to the beginning of initial treatment. The recruitment will be carried out with a sample at convenience in patients with brain tumors in terminal phase that are outside conventional treatment. The therapy with quantum magnetic resonance (Cytotron®) will be administered as a compassionate treatment with the authorization signed by the parents and with the respective informed consent (depending on age).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QMRT using the Cytotron® (Experimental): Experimental: QMRT using the Cytotron® Intervention: 28 days of treatment with QMRT with the Cytotron®. Patients diagnosed with terminal brain tumors between 3 and 16 years of age whose parents agree to participate in the study and have signed informed consent and informed consent in patients with age or mental age over 8 years.
  Interventions: Procedure: QMRT with the Cytotron®

INTERVENTIONS:
Procedure: QMRT with the Cytotron® — Cytotron® utilizes a combination of instantaneous magnetic field and RF at the safe, lowerend of the EM spectrum. Radiofrequency waves are computed based on individualized PD measurements of the target lesion(s) for therapeutic purpose. Its working principle is based on the underlying theory of magnetic resonance.
  Other Names: Rotational Field Quantum Magnetic Resonance (RFQMR) Technology platform

SUMMARY:
This is a prospective case-control study. This study is expected to last for approximately 12 months, comprised of 4-8 weeks of enrollment period, 28 days of treatment and 6 months of follow up. The enrollment will be completed prior to the beginning of initial treatment. The study will be closed when 10 subjects have completed the study. The recruitment will be carried out with a sample at convenience.

DETAILED DESCRIPTION:
A case-study study. The controls will be historical and matched to the age range (preschool, school age, early adolescent, late adolescent) and type of tumor. This study is expected to last for approximately 12 months, comprised of 4-8 weeks of enrollment period, 28 days of treatment and 6 months of follow up. The recruitment will be carried out with a sample at convenience in patients with brain tumors in terminal phase that are outside conventional treatment. Quantum magnetic resonance therapy (QMRT) will be administrated with the Cytotron® device.. The CYTOTRON-RTE-6040-864GEN (Class IIA Medical Therapeutic Device; developed by Scalene Cybernetics Ltd, Bengaluru, India), is a patented (U.S. Patent 9162076 B2 awarded 20/10 2015, European Patent EP 175350831, awarded 3/11/2015, Chinese Patent issued 2010, 09/08), CE marked device. QMRT will be administered as a compassionate treatment with the authorization signed by the parent(s) and with the respective informed consent (depending on age). Study Center: Hospital Infantil de México Federico Gómez. Objectives: To determine the safety and efficacy of QMRT using the Cytotron in terminal brain tumors. Number of Subjects: 10. Diagnosis and main Inclusion Criteria Subjects with clinically diagnosed terminal brain tumors, age: 3 to 16. Study Device, Dose,Route Device: Cytotron-generated precisely computed, individualized Dosimetry with Radiofrequencies (RF) in the presence of a pulsed, instantaneous electromagnetic resonance (MR) field, applied to a subject. Dose: 1 hour per day. Route: Focused, non-invasive RF and MR beams delivered to target areas identified by brain MRI scan and individual proton density (PD) measurements of the target lesions. Duration of administration: Once a day for 28 consecutive days. Reference therapy: None

ELIGIBILITY:
Inclusion Criteria:

* A child 3 to 16 years of age.
* A clinical diagnosis of terminal primary brain tumor
* A diagnosis of a terminal brain tumor, which indicates that the patient is out of conventional treatment and does not have another therapeutic option.

Exclusion Criteria:

* Patients with metastasis
* Patients requiring oxygen or mechanical ventilation
* Current or recent history (within 2 months) of significant bacterial, fungal, viral, or mycobacterial infection.
* Having a condition considered as causing or likely to cause co-morbidities, as determined by the investigator based on medical history, physical examination, vital signs, and clinical laboratory tests.
* Subject with magnetic implants, pacemakers, claustrophobia or any other condition that precludes them from entering or staying in the treatment device.
* Children with previous neurosurgery within 6 months at the time of screening.
* History of myocardial infarction, congestive heart failure, or stroke.
* Subject is exposed to secondary smoking in his/her home environment.
* Subjects who are unable or unlikely to comply with the protocol, determined by the majority vote of the investigators.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life with the Pediatric Quality of Life Inventory (PedsQL) brain tumors | 6 months
  Change in the total score in the PedsQL of the patients diagnosed with brain tumor will be measured before starting the treatment and 6 months later. Higher values are going to represent a better outcome.

SECONDARY OUTCOMES:
Measuring the increase, decrease, or change in the use of medication use for seizure or spasticity | 6 months
  The change in the use of medications use for seizure or spasticity as a symptom manifestation in children brain tumors before initiating the treatment and 6 months later will be measured.
Measuring the change in the number of seizures during the study period. | 6 months
  The change in the use of the number of epileptic seizures of the patients diagnosed with terminal brain tumor before initiating the treatment and 6 months later will be measured.
Change of brain activities using fMRI | 6 month
  Identifying the change in representative modules, visual, motor and basal ganglia measuring the brain activities during resting state before and after treatment.
Change of brain activities using the Diffusion tensor imaging in MRI | 6 month
  Identifying the change in representative modules, visual, motor and basal ganglia by measuring diffusion tensor data and the anisotropic diffusion of the brain before and after treatment.
Change of brain activities using the EEG. | 6 month
  Identifying the change in electrical activity in the brain before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Juan C García Beristain, MD, Study Director — Hospital Infantil de Mexico Federico Gomez
Locations (1):
- Hospital infantil de México Federico Gomez, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barragan-Perez EJ, Alvarez-Amado DE, Dies-Suarez P, Tobon SH, Garcia-Beristain JC, Penaloza-Gonzalez JG. Compassionate use of Quantum Magnetic Resonance Therapy for treatment of children with Diffuse Brainstem Glioma in Mexico City: a single institutional experience. J Neurooncol. 2022 Apr;157(2):377-382. doi: 10.1007/s11060-022-03972-2. Epub 2022 Mar 10. PMID 35266065